CLINICAL TRIAL: NCT06984380
Title: Tele-Rehabilitation Intervention in Community-Based Healthcare for Patients With Osteoporosis (DHEAL-COM-OP)
Acronym: DHEAL-COM-OP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: INRCA_006_2024
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Osteoporosis; Older People
MeSH Terms: conditions — Osteoporosis | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Older patients with osteoporosis
  Interventions: Other: Telerehabilitation
- Usual care (Sham Comparator): Older patients with osteoporosis
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Telerehabilitation — Patients will receive a personalised home tele-rehabilitation exercise program consisting of 3 sessions per week for a duration of 12 weeks. BTS TELEREHAB is a platform that allows the delivery of remote rehabilitation services. The patient is given the system to take home, where they will connect the small Brain PC, that is the computer unit of the BTS TELEREHAB solution, to their television. During motor rehabilitation sessions, the patient wears a special inertial sensor, the G-Sensor device, that measures movements in real-time, allowing the clinician to remotely monitor the correct execution of the exercises. In addition to the proposed therapeutic exercises, functional assessment tests are also included for patient follow-up. The presence of the inertial sensor supports the clinician in verifying the correct execution of the motor task and in the precise quantification of joint mobility.
  Arms: Intervention arm
Other: Usual care — Participants will receive a booklet containing information and activities on well- being. They will be invited to do whatever they wish with the information booklet and the proposed exercises.
  Arms: Usual care

SUMMARY:
The DHEAL-COM-OP study is characterized as a feasibility study. The general objective is to evaluate the improvement in the physical performance of patients with osteoporosis detected through the Performance-Oriented Mobility Assessment (POMA) scale, following a rehabilitation intervention integrated with the BTS TELEREHAB technology.

DETAILED DESCRIPTION:
The DHEAL COM project aims to evaluate the improvement in physical performance of patients with osteoporosis following a rehabilitation intervention integrated with technology in telerehabilitation. Specifically, the project aims to develop a telerehabilitation platform that enables people to perform physical activity at home.

The first objective of the project is to evaluate the improvement of physical performance, in terms of gait and balance capability, of patients with osteoporosis detected through the Tinetti Performance Oriented Mobility Assessment (POMA) scale following an integrated rehabilitation intervention with BTS TELEREHAB technology.

Forty elderly people with osteoporosis aged at least 65 years who wish to participate in the study and who meet the inclusion and exclusion criteria. Participants will be randomized into experimental group (GS) and control group (GC). Patients in the experimental group will receive a personalized program of home tele-rehabilitation exercises divided into 3 workouts per week, for a duration of 12 weeks. The training sessions will be organized as follows: one session will be carried out in telerehabilitation with the support of the physiotherapist in small groups of maximum 5 patients; in the remaining two the patient will perform the exercises independently at home. Before starting the rehabilitation program, the patient will receive training with the technology in the hospital, in the presence of the physiotherapist.

Patients in the control group will be offered activities to perform at home, with the same frequency, in line with the usual care activities already proposed by the Rehabilitation Unit.

Patients will be contacted periodically by the physiotherapist to evaluate the improvement of the main and secondary outcomes detailed in the following protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a positive MOC for osteoporosis without a history of major fractures (femur and vertebrae);
* Functional Ambulation Category (FAC) score ≥ 3;
* Stability of drug treatment for at least 1 month;
* Maintaining an upright position independently > 30";
* Mini-Mental State Examination (MMSE) ≥ 24;
* Geriatric depression scale (GDS) < 2;

Exclusion Criteria:

* Myocardial infarction or stroke within 6 months;
* Painful arthritis, spinal stenosis, amputation, painful foot lesions, or neuropathy that limits balance and mobility;
* Uncontrolled hypertension
* Metastatic cancer or immunosuppressive therapy;
* Significant visual or hearing impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in physical performance | At baseline and 12 weeks later
  The physical performance, in terms of balance and gait ability, will be detected through the Tinetti Performance Oriented Mobility Assessment (POMA) scale. The maximum possible score is 28 points. The total POMA score provides an indication of an individual's fall risk:
  * 25-28 points: Indicates a low risk of falls
  * 19-24 points: Indicates a medium or moderate risk of falls
  * Less than 19 points (< 19): Indicates a high risk of falls
  The improvement is assessed in an increase in the POMA score of at least 3 points.

SECONDARY OUTCOMES:
Improvement in physical function | At baseline and 12 weeks later
  Physical performance will be assessed using the Short Physical Performance Battery (SPPB). The total SPPB score ranges from 0 to 12, with 12 indicating the best performance.
Improvement in quality of life | At baseline and 12 weeks later
  The quality of life will be evaluated by the SF-12 Health Survey (SF-12). It consists of 12 items that produce two measures related to two different aspects of health: physical health (PCS) and mental health (MCS). Both typically ranging from 0 to 100, where 0 represents the worst health status and 100 represents the best health status.
Improvement in mobility | At baseline and 12 weeks later
  The mobility will be measured by the Time Up and Go (TUG) test. It measures the time it takes a person to get up from a chair, walk three meters, turn around, return to the chair, and sit down again. During the test, the person should wear regularly used shoes and use any normally used Mobility Aids. A score of ten seconds or less indicates normal mobility; times between 11 and 20 seconds are within normal limits for frail elderly and disabled patients; times greater than 20 seconds indicate that the person needs outside assistance and the need for further examination and intervention. A score above 30 seconds suggests that the person may be prone to falls

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Renato Riccardi, MD, Study Director — IRCCS INRCA, Ancona, Italy
Locations (1):
- IRCCS INRCA Hospital, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No